CLINICAL TRIAL: NCT04149548
Title: Placental Assessment in Early and Late Pregnancy in Diabetic Women
Brief Title: Placental Assessment in Diabetic Mothers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Researcher ,National research centre and Algezeera hospital, Aljazeera Hospital
Other Study IDs: Diabetes mellitus
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant diabetic women: Fetal Ultrasound to diabetic pregnant women
  Interventions: Diagnostic Test: ultrasound
- non diabetic pregnant women: Fetal ultrasound to non diabetic pregnant women
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — Obstetric ultrasound to pregnant women

SUMMARY:
Diabetes mellitus is one of the major heath problems

DETAILED DESCRIPTION:
Maternal and fetal effects are edpected to be more than in diabetic mothers

ELIGIBILITY:
Inclusion Criteria:

* in control group A non diabetic pregnant women

Exclusion Criteria:

* Diabetic pregnant women

And the reverse in group B

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Diabetic and non diabetic pregnanrt women attending for ANC
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-11-06 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
The number of diabetic fetuses who will have undesirable effects | within 6 months
  Number of fetuses with macrosomia and other diabetes effects

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — Algezeera
Locations (2):
- Egypt (2):
  - Algazeerah and Kasralainy hospital, Giza
  - Algazeerah, Giza